CLINICAL TRIAL: NCT02894424
Title: Pilot Study of the Effect on the Retinal Sensitivity of the Membrane Blue Dual® Dye Used for Peeling of the Internal Limiting Membrane in Macular Hole Surgery
Brief Title: Effect of the Membrane Blue Dual® Dye on the Retinal Sensitivity in Macular Hole Surgery
Acronym: MICROCOL
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: YLR_2015_4
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Macular Hole Surgery
Keywords: Inner limiting membrane; Microperimetry; surgical's dye

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The idiopathic macular hole, age-related disease, is a major cause of vision loss and affects at least two persons in 1000 after 40 years.

This hole causes an acute decline linked to a central scotoma. The only treatment is surgical. The surgery involves removing the posterior hyaloid (vitreous base) to relieve the tensile forces. To be sure the removed is complete and to facilitate the closure of the hole, a peeling of the internal limiting, the outermost layer of the retina, is often suggested. The inner limiting membrane (ILM), transparent and adherent to the retina, is colored with vital dyes to facilitate its removal. After closure of the macular hole, the central scotoma disappears but a diffuse and asymptomatic loss of pericentral sensitivity is often described. This sensitivity decrease could be induced by the dyes used during surgery.

This effect has not been studied clinically for recent dyes (Membrane Blue Dual®, Brilliant Blue®, Acid Violet®) at the concentrations used, but is known in electrophysiology at higher concentrations, at least on the isolated retina models.

It would be interesting to search for a decrease in retinal peri-foveal postoperative sensitivity after surgery of macular holes, performed with the usual dyes. Only microperimetry can observe this decrease in retinal sensitivity. This is a noninvasive technique that explores the macular visual field. It is performed without iris dilatation and allows an automatic exploration ensuring rapid and accurate analysis of retinal sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* lower idiopathic macular hole inferior or equal to 600 micron millimeter
* undergoing macular hole surgery

Exclusion Criteria:

* Myopia > -3 diopters
* pregnant women
* no Health Insurance coverage
* refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred for macular hole surgery
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2017-02-23 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-10-05 (Actual)

PRIMARY OUTCOMES:
change in retinal sensitivity | change from baseline sensitivity at 1 month after macular hole surgery
  change from baseline sensitivity at 1 month after macular hole surgery

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Le Mer, MD, Principal Investigator — Fondation OPH A de Rothschild
Locations (2):
- France (2):
  - CHU Dijon, Dijon
  - Fondation Ophtalmologique A. de Rotchschild, Paris